CLINICAL TRIAL: NCT06389331
Title: A Comparative Study on Effects of Defect Closure Versus Non-Closure in Laparoscopic Totally Extraperitoneal Repair of Direct Inguinal Hernia
Brief Title: Study on Effects of Defect Closure in Laparoscopic Repair of Direct Inguinal Hernia
Status: Completed | Type: Observational
Sponsor: B.P. Koirala Institute of Health Sciences (Other)
Responsible Party: Principal Investigator, Vijay Pratap Sah, doctor, B.P. Koirala Institute of Health Sciences
Other Study IDs: IRC/1971/020
Record Dates: First submitted 2024-04-24; First posted 2024-04-29 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Hernia; Direct Inguinal Hernia; Seroma Following Procedure
Keywords: TEP; Direct Hernia Closure; Seroma Formation; Pain
MeSH Terms: conditions — Hernia; Hernia, Inguinal; Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- defect closure: the fascia transversalis (pseudo sac) was pulled and incorporated into closure with a non-absorbable polypropylene barbed monofilament size-0 suture
  Interventions: Other: closed the defect with barbed suture
- non closure group: defect was left open

INTERVENTIONS:
Other: closed the defect with barbed suture — In direct hernia, content was reduced, and the fascia transversalis (pseudo sac) was pulled and incorporated into closure with a non-absorbable polypropylene barbed monofilament size-0 suture
  Groups: defect closure

SUMMARY:
The defect closure was found to have higher pain and less seroma formation at various intervals of time following TEP for moderate-large direct inguinal hernia. Although these findings were statistically insignificant, they may be clinically significant, and further studies with a larger sample size are suggested.

DETAILED DESCRIPTION:
Inguinal hernia is a common and widespread condition from which millions of people suffer. Repair of an inguinal hernia is one of the most frequently performed operations in general surgery. Totally extraperitoneal (TEP) and transabdominal preperitoneal (TAPP) repair are the principal techniques in laparoscopic hernia repair. Laparoscopic hernia repair is recommended for bilateral and recurrent inguinal hernias. It has also been recommended for patients with primary unilateral inguinal hernia, contingent on the availability of surgical expertise and resources, due to a lower incidence of post-operative pain and chronic pain.

Seroma formation is a frequent complication of laparoscopic mesh repair of moderate-large direct inguinal hernia defects. While rates of seroma formation have been reported to be as high as 10-30%. Several attempts have been made to reduce the incidence of seroma formation, such as tacking the transversalis fascia (TF) to the ramus of the pubis, closing the direct inguinal hernia defect via the endoloop technique, and filling the potential dead space with fibrin glue. However, there is a potential increase in the risk of infection and also a risk of chronic pubic bone pain from the tack staples or vasculo-nervous injury if fixing the TF to the abdominal wall, which would lead to extra discomfort for the patient. The closure of a direct hernia defect with a barbed suture not only closes the defect superficially but also exterminates the defect cavity; consequently, the incidence of seroma formation has been greatly reduced.

However, there is still controversial evidence regarding the choice of the two procedures in terms of reducing the rate of seroma formation and pain. Thus, it is ambiguous which surgical technique should be considered best to repair an inguinal hernia. In this study, we tried to evaluate the technical aspect of direct defect closure in laparoscopic TEP inguinal hernia repair and its effect on the primary outcomes in terms of seroma formation and pain at different time intervals, along with the secondary outcomes such as operative time, length of postoperative hospital stay, days to resume normal activities, recurrence, and intraoperative complications like injury to the vas, vessel, and visceral injury or peritoneal tear.

ELIGIBILITY:
Inclusion Criteria:

* age greater than 18 years
* uncomplicated direct inguinal hernia (≥M3)

Exclusion Criteria:

* defect size ≤M2
* complicated hernia (irreducible, obstructed, or recurrent hernia)
* patients unfit for general anesthesia

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with inguinal hernia presenting to surgery OPD
Sampling Method: Probability Sample
Enrollment: 88 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
seroma formation in defect closure group | till 6 months
  After closing the defect, there is less seroma formation than in the defect non closure group

CONTACTS AND LOCATIONS:
Overall Officials: Rakesh Kumar Gupta, MS, Principal Investigator — B. P. Koirala institute of health science
Locations (1):
- Vijay Pratap Sah, Malaṅgawā, Madhesh Pradesh, Nepal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rutkow IM, Robbins AW. Demographic, classificatory, and socioeconomic aspects of hernia repair in the United States. Surg Clin North Am. 1993 Jun;73(3):413-26. doi: 10.1016/s0039-6109(16)46027-5. PMID 8497793
- [Background] McKernan JB, Laws HL. Laparoscopic repair of inguinal hernias using a totally extraperitoneal prosthetic approach. Surg Endosc. 1993 Jan-Feb;7(1):26-8. doi: 10.1007/BF00591232. PMID 8424228
- [Background] Usmani F, Wijerathne S, Malik S, Yeo C, Rao J, Lomanto D. Effect of direct defect closure during laparoscopic inguinal hernia repair ("TEP/TAPP plus" technique) on post-operative outcomes. Hernia. 2020 Feb;24(1):167-171. doi: 10.1007/s10029-019-02036-1. Epub 2019 Sep 6. PMID 31493054
- [Background] Kockerling F, Bittner R, Adolf D, Fortelny R, Niebuhr H, Mayer F, Schug-Pass C. Seroma following transabdominal preperitoneal patch plasty (TAPP): incidence, risk factors, and preventive measures. Surg Endosc. 2018 May;32(5):2222-2231. doi: 10.1007/s00464-017-5912-3. Epub 2017 Oct 26. PMID 29075973

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2020-09-01): https://cdn.clinicaltrials.gov/large-docs/31/NCT06389331/Prot_ICF_000.pdf